CLINICAL TRIAL: NCT02889146
Title: Using a Progressive Mobility Program and Technology to Increase the Level of Physical Activity and Its Benefits in Respiratory, Muscular System and Functionality of ICU Patients: a Randomized Clinical Trial
Brief Title: Progressive Mobility Program and Technology to Improve the Level of Physical Activity and Functionality of ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: deborass
Record Dates: First submitted 2016-03-03; First posted 2016-09-05 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Critical Illness; Muscle Weakness
Keywords: Intensive Care Units; Physical Therapy Specialty; Critical illness; Muscle weakness; Bed rest
MeSH Terms: conditions — Critical Illness; Muscle Weakness | interventions — Respiratory Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional Physical Therapy: motor physical therapy delivered by the intensive care unit physical therapists, according to his own criteria, without following any protocol. Respiratory therapy.
  Interventions: Other: Conventional Physical Therapy; Other: Respiratory therapy
- Protocol group (Experimental): Early and progressive mobilization program: motor physical therapy delivered by a trained physical therapist according to the mobilization protocol, in which patient progress according to his performance. Respiratory therapy.
  Interventions: Other: Early and progressive mobilization program; Other: Respiratory therapy

INTERVENTIONS:
Other: Conventional Physical Therapy — Control group will receive respiratory therapy according to the service routine and conventional physical therapy. Conventional physical therapy will be offered by the hospital physical therapists, according to their own criteria. Consists of passive, assisted and resisted mobilization, positioning in bed, transferring to bedside or chair, orthostatism and deambulation, however without a definition of a protocol. The physical therapist will be responsible for the choice of the techniques employed in each session. There will be no previous definition of the next sessions. No technology equipment will be used in this group, since they are not available in the routine care.
  Arms: Control group
Other: Early and progressive mobilization program — Protocol group will receive respiratory therapy according to the service routine and motor physical therapy according to the program of early and progressive mobilization. Patients will receive the program once daily during the intensive care unit stay, offered by a trained physical therapist, at the adequate level according to the level of consciousness and muscle strength. The program contains by techniques for muscle length and muscle strength maintenance or gain, aerobic exercises, exercises for gait rehabilitation and cognitive components. Patient will progress to the next level of the protocol completing the previous level. Technology equipment available: functional electrical stimulation device, dumbbells, cycle ergometer, fixed walker, ambulation assistive device and video game.
  Arms: Protocol group
Other: Respiratory therapy — Respiratory therapy according to the service routine.

SUMMARY:
The purpose of this study is to verify if a protocol of early and progressive mobility which includes the use of technology is able to increase the level of physical activity and improve functionality and respiratory and muscular function of Intensive Care Unit patients compared with conventional Physical Therapy.

DETAILED DESCRIPTION:
The evolution of treatment in the Intensive Care Unit (ICU) has increased the survival and morbidity post hospital. Functional disability in these patients has its main factor in the weakness and loss of muscle mass, which is the major complications reported by these patients. The most negative result in long-term post ICU is the impact on quality of life and functional decline due to muscle disorders and fitness. This is achieved by the period of inactivity and prolonged rest, leading to losses and changes in various body systems. Given these facts, interventions for greater mobility in bed and out of it are very important. Early mobility programs has proved beneficial, however, as in other types of rehabilitation, the exercises should be prescribed with its specific characteristics, including the intensity. However, little has been described in the researches abut the activity level in the ICU, and using a quantitative measure. The use of technology seems to facilitate the offering of this type of therapy, supplying the limitations. Therefore, there are little evidences about these topics and randomized controlled studies to investigate these factors.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the Emergency Intensive Care Unit of Clinical Hospital, Medical School, University os Sao Paulo
* inspired oxygen fraction ≤ 60%
* positive end expiratory pressure ≤ 10 points
* peripheral oxygen saturation ≥ 90%
* respiratory rate ≤ 35
* without cardiac arrhythmia or acute ischaemia
* heart rate > 50 bpm and < 140 bpm
* without high or raising dose of vasoactive drugs
* mean body pressure > 60 mmHg and < 120 mmHg
* without active bleeding
* without prescribed bedrest

Exclusion Criteria:

* transference from other hospital
* diagnosis of neurological disorders
* intensive care unit stay < 4 days
* contraindication to mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Functional status | At the time of discharge from the ICU, at least 4 days after admission.
  Ability to perform daily living activities assessed by Barthel Index

SECONDARY OUTCOMES:
Level of physical activity during the whole intensive care unit stay | At the time of discharge from the ICU, at least 4 days after admission.
  Level of physical activity measured by an accelerometer
Pulmonary function | At the time of discharge from the ICU, at least 4 days after admission.
  Pulmonary function assessed by a spirometer
Maximum inspiratory pressure | At the time of discharge from the ICU, at least 4 days after admission.
  Maximum inspiratory pressure measured by an specific equipment
Peripheral muscle strength | At the time of discharge from the ICU, at least 4 days after admission.
  Muscle strength assessed by hand grip dynamometer
Electromyography muscle activity | At the time of discharge from the ICU, at least 4 days after admission.
  Quadriceps femoris electric activity assessed by surface electromyography
Muscle function and mobility | At the time of discharge from the ICU, at least 4 days after admission.
  Test by Time up and Go
Intensive care unit length of stay | At the time of discharge from the ICU, at least 4 days after admission.
  Count of the number of days spent at the intensive care unit
Correlation between physiological variables and the level of physical activity | At the time of discharge from the ICU, at least 4 days after admission.
  Correlation between the physiological variables collected during the study and the level of physical activity measured by the accelerometer
ICU mobility Scale | Through study completion, an average of 2 weeks
  Measure of mobility milestones in critically ill patients.
Long term follow up | After three months and one year of discharge
  Longer-term follow-up for functional status by Barthel Index after three months and one year of discharge
Level of activity by Perceived Exertion | approximately 40 minutes after therapy, immediately after the end of the protocol
  Level of exercise by Perceived Exertion by Borg Rating of Perceived Exertion Scale

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fu, PhD, Principal Investigator — Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy - Medical School of University of Sao Paulo
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy - Medical School of University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gomes TT, Schujmann DS, Fu C. Rehabilitation through virtual reality: physical activity of patients admitted to the intensive care unit. Rev Bras Ter Intensiva. 2019 Oct-Dec;31(4):456-463. doi: 10.5935/0103-507X.20190078. PMID 31967219
- [Derived] Schujmann DS, Lunardi AC, Fu C. Progressive mobility program and technology to increase the level of physical activity and its benefits in respiratory, muscular system, and functionality of ICU patients: study protocol for a randomized controlled trial. Trials. 2018 May 10;19(1):274. doi: 10.1186/s13063-018-2641-4. PMID 29747662